CLINICAL TRIAL: NCT02233348
Title: Neurocognitive and Psychosocial Outcome of Youths With Autism Spectrum Disorder: a Follow-up Study
Brief Title: Neurocognitive and Psychosocial Outcome of Youths With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201403109RINC
Record Dates: First submitted 2014-08-27; First posted 2014-09-08 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ASD group: Subjects with DSM-IV ASD diagnosis
- Control group: Controls without lifetime ASD or a family history of ASD

SUMMARY:
Autism spectrum disorders (ASD) is a common childhood-onset, multi-factorial, highly heritable, clinically and genetically heterogeneous, neurodevelopmental disorder. Due to its high prevalence and severe lifelong impairment without effective prevention and treatment, there is a dearth of investigating its pathogenesis, longitudinal outcome, and biomarkers (endophenotypes). The ultimate goals of this 5-year project are to prospectively investigate the outcome and changes of psychosocial and neurocognitive functions of a cohort of probands with ASD at adolescence and young adulthood as the primary aim; and to test whether structural and functional brain connectivity can be effective endophenotypes of ASD using the unaffected sibling and follow-up designs as the secondary aims.

DETAILED DESCRIPTION:
Primary Aim:

To investigate the neuropsychological, neuroimaging, social cognitive, and psychosocial outcomes at adolescence and young adulthood among children with ASD as compared to typically developing (TD) controls.

Secondary Aims:

1. To examine the changes and stability of ASD core symptoms, neuropsychological function, structured and functional connectivity, psychosocial functions over a 4-7 year follow-up period.
2. To identify early individual (clinical, behavioral, and neurocognitive variables), family, school, environmental factors to predict the neurocognitive and psychosocial outcomes at adolescence and young adulthood.
3. To validate the neuropsychological functioning (e.g., set-shifting, executive function, and visuo-spatial memory etc.) and structural (morphometric,, cortical thickness, gyrification, white matter tract integrity) and functional connectivity (resting-state and social task fMRI) in fronto-temporal, cortico-striato-thalamic, default mode network, and other circuits as effective imaging endophenotypes (biomarkers) by demonstrating the stability of these imaging data and the intermediate position of unaffected siblings between ASD probands and age-, sex-, handedness-, and IQ-matched TD at Time 1 and follow-up.
4. To correlate the data from structural and functional connectivity, neuropsychology and ASD core symptoms stratifying by proband-unaffected sibling dyads, and different developmental stages.
5. To collect blood sample, and to analyze neurodevelopmental and immune genes, cytokine level, and environmental exposure.

ELIGIBILITY:
Inclusion Criteria:

ASD participants

1. that they have a clinical diagnosis of autistic disorder or Asperger disorder defined by the DSM-IV and ICD-10 criteria, made by board-certificated child psychiatrists and who were clinically diagnosed with ASD confirmed by the ADI-R 7 years ago;
2. their ages range from 10 to 25 (i.e., 3-18 years old at the first assessment);
3. both parents are Han Chinese;
4. who have complete clinical and behavioral data at the 1st assessment;
5. participants and their parents consented to participate in this longitudinal study 7 years ago for complete assessments (3 visits of assessments) at follow-up.

Inclusion Criteria for TD controls, who will be recruited either by school teachers or from the community, are that they are Han Chinese, consent to the study (if age <18, parents, too) to complete all the assessments.

Exclusion Criteria:

For TD controls:

1. comorbidity with DSM-IV-TR or DSM-5 diagnoses of ASD, ADHD, schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorder, organic psychosis, schizotypal personality disorder, bipolar disorder, depression, severe anxiety disorders or substance use;
2. comorbidity with neurological or systemic disorders; and
3. having a first degree relative who may have ASD based on family history method assessment.

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 373 ASD, aged 10-25, from the cohort of ASD established by NRPGM, who consented to this follow-up study at their first assessments in 2007-2011 and 150 age-, and sex-matched TD, at the ratio of 2:1.
Sampling Method: Non-Probability Sample
Enrollment: 523 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of autism | one day
  Using Autism Diagnostic Interview-Revised (ADI-R) to assess the developmental and behavioral aspects of autism, including reciprocal social interaction, communication, and repetitive behaviors and stereotyped patterns.

SECONDARY OUTCOMES:
Diagnosis of autism | one day
  Using Autism Diagnostic Observation Scale (ADOS) to assess social communication, social relatedness, play, imaginative of materials, and restricted and/or repetitive behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan